CLINICAL TRIAL: NCT01274507
Title: A Multicenter Longitudinal Study for Disease Profiling of Asthma and Chronic Obstructive Pulmonary Disease
Brief Title: A Study for Disease Profiling of Asthma and Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR017362; NOCOMPOUNDASH0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-10-28; First posted 2011-01-11 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2014-09

CONDITIONS: Asthma; Pulmonary Disease, Chronic Obstructive
Keywords: Asthma; Pulmonary Disease, Chronic Obstructive; Healthy; Longitudinal Study; Bronchoscopy
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Other)
  Interventions: Other: Medical tests

INTERVENTIONS:
Other: Medical tests — All participants will undergo medical tests and will be observed.

SUMMARY:
The purpose of this study is to characterize the clinical, physiologic, and molecular profiles of healthy participants, participants with mild, moderate, and severe asthma; and participants with moderate to severe Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is a multi-center, longitudinal (participants are followed over long period of time with continuous or repeated observations of health outcomes) exploratory study (biomarkers, clinical and physiological parameters for participants with asthma and COPD are observed for the first time). This study will be conducted in 2 parts. Part 1 will include healthy participants and participants with mild, moderate, and severe asthma. Part 2 will include healthy nonsmokers, healthy asymptomatic smokers, and participants with moderate and or severe COPD. Study participants will undergo medical tests that will include pulmonary function testing, assessment of airway reactivity, bronchoscopy procedure, blood samples for routine laboratory tests, biomarkers and DNA evaluation (for some study participants), induced sputum collection, and exhaled nitric oxide collection. Safety evaluations will includes assessment of adverse events, clinical laboratory tests, 12-lead electrocardiogram, vital signs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Age: for Part 1, healthy: 18 and 55 years; for Part 1, asthma: 18 and 70 years; for Part 2, nonsmokers: 40 and 65 years; for Part 2, smokers: 40 and 65 years; for Part 2, chronic obstructive pulmonary disease (COPD): 40 and 65 years
* Having mild, moderate, or severe asthma (for Part 1, asthma)
* Clinically stable asthma and have been on their current asthma controller therapy for at least 6 weeks prior to screening (for Part 1, asthma)
* No history of chronic respiratory disease including asthma (for Part 2, nonsmokers)
* Be a nonsmoker for 1 year or more at initial screening visit and have 10 packs or less per year history of smoking (for all Part 1 and Pat 2, nonsmokers)
* Be a current smoker with a current history of at least 20 pack years (for Part 2, smokers)
* Stable COPD in the 3 months prior to screening (for Part 2, COPD)
* Treating with Beta-adrenergic receptor agonist, anticholinergic bronchodilators, inhaled corticosteroid at stable doses for at least 4 weeks prior to screening (for Part 2, COPD)

Exclusion Criteria:

* History of sleep apnea requiring medical intervention and positive urine pregnancy screening result (for all Part 1 and Part 2)
* Positive urine screen for nicotine; positive serology test for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, or hepatitis C virus antibody at screening (for all Part 1 and Part 2)
* Allergic bronchopulmonary aspergillosis, allergic bronchopulmonary mycosis, or occupational asthma (for Part 1, asthma)
* Requires long term oxygen therapy on a daily basis for chronic hypoxemia at screening visit except when used for exercise only (for Part 2, COPD)
* Pneumonia, COPD exacerbation that required systemic steroids, upper or lower respiratory tract infection, lung cancer surgery, lung volume reduction, or a lung transplant (for Part 2, COPD)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaire (AQLQ) score | Baseline (5 to 14 days after screening), Month 3, Month 6, and Month 12 (for Part 1: participants with asthma)
  AQLQ is used to measure the physical, emotional, social and occupational problems for participants with asthma. There are 32 questions in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli) to measure activity limitation and symptom frequency using a recall period of 2 weeks. Each 32 questions are on a 7-point scale (7 = not impaired at all and 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains. Lower scores indicate worsening.
Asthma Control Questionnaire (ACQ) score | Baseline, Month 3, Month 6, and Month 12 (for Part 1: participants with asthma)
  ACQ is used to evaluate asthma control, the full range of clinical impairment (well controlled to life threatening) for the participant with asthma. There are 7 questions (5 for symptoms [night-time awakenings, morning symptoms, limitation of activities, shortness of breath, and wheezing], use of daily rescue bronchodilator, and percent predicted forced expiratory volume value). All 7 items are scored on a 7-point scale (0 = good control, 6 = poor control), with the mean score as an overall summary score. The recall period is 7 days. Higher scores indicate worsening.
Forced Expiratory Volume in 1 second (FEV1) value | Screening, Baseline, 5 to 14 days after baseline (for Part 1: healthy participants); and Month 3, Month 6, and Month 12 (for Part 1: participants with asthma and for all Part 2 participants)
  FEV1 will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the volume and/or flow of air that can be inhaled and exhaled. Lung volumes will be measured according to the body temperature, pressure, and saturated standard convention using the spirometer. Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol and post- bronchodilator spirometry will be performed after 15 to 30 minutes administration of albuterol/salbutamol via metered-dose inhaler.
Forced Vital Capacity (FVC) value | Screening, Baseline, 5 to 14 days after baseline (for Part 1: healthy participants); and Month 3, Month 6, and Month 12 (for Part 1: participants with asthma and for all Part 2 participants)
  FVC will be measured by using spirometry test. Spirometry is used to measure lung function, specifically the volume and/or flow of air that can be inhaled and exhaled. Lung volumes will be measured according to the body temperature, pressure, and saturated standard convention using the spirometer. Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol and post- bronchodilator spirometry will be performed after 15 to 30 minutes administration of albuterol/salbutamol via metered-dose inhaler.
Forced Expiratory Flow (FEF) 25-75 value | Screening, Baseline, 5 to 14 days after baseline (for Part 1: healthy participants); and Month 3, Month 6, and Month 12 (for Part 1: participants with asthma and for all Part 2 participants)
  FEF is the flow of air coming out of the lung during the middle portion of a forced expiration. It is generally defined by what fraction remains of the forced vital capacity (FVC), usually 25-75 percent (FEF25-75%). Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol and post- bronchodilator spirometry will be performed after 15 to 30 minutes administration of albuterol/salbutamol via metered-dose inhaler.
Peak Expiratory Flow Rate (PEFR) | Screening, Baseline, 5 to 14 days after baseline (for Part 1: healthy participants); and Month 3, Month 6, and Month 12 (for Part 1: participants with asthma and for all Part 2 participants)
  PEER will be measures by using spirometry test. Spirometry is used to measure lung function, specifically the volume and/or flow of air that can be inhaled and exhaled. Lung volumes will be measured according to the body temperature, pressure, and saturated standard convention using the spirometer. Pre-bronchodilator spirometry will be performed in the absence of albuterol/salbutamol or at least 6 hours after the last dose of albuterol/salbutamol and post- bronchodilator spirometry will be performed after 15 to 30 minutes administration of albuterol/salbutamol via metered-dose inhaler.
Methacholine challenge | Screening or Baseline (for Part 1: participants with asthma)
  Methacholine challenge test is used to assess airway reactivity in asthma. In this test, baseline spirometry for participant is measured by inhalation of increasing concentrations of aerosolized methacholine up to 16 mg/mL. The provocative dose (PC20) is defined as the dose of methacholine required to cause a greater than or equal to 20 percent decrease from the baseline forced expiratory volume in 1 second value. A PC20 result of less than or equal to 16 mg/mL will be considered to reflect increase airway responsiveness for fulfilling eligibility criteria.
Fractional Exhaled Nitric Oxide (FENO) | Baseline, Month 3, Month 6, and Month 12 (for Part 1: participants with asthma); and 5 to 14 days after baseline (for Part 2: participants with chronic obstructive pulmonary disease)
  Measurement of FENO is a quantitative, noninvasive, simple, and safe method of measuring airway inflammation that provides a complementary tool to assessing airways disease. The participant can exhale directly into a measurement device, or into a reservoir that can afterwards be connected to the analyzer. With the former technique, the early and later nitric oxide in the breath sample can be analyzed separately. Two replicate FENO measurements will be obtained that agree at the 10% level and up to a total of 8 measurements will be performed to achieve this level of agreement.
Induced sputum | Screening, Baseline (for Part 1: healthy participants and for all Part 2 participants); and Month 6 (for Part 1: participants with asthma)
Saint George's Respiratory Questionnaire score for Chronic Obstructive Pulmonary Disease (COPD) participants (SGRQ-C) | Baseline (for Part 2: participants with COPD)
  SGRQ-C is a 14-item questionnaire designed to measure health impairment in participants with COPD. The SGRQ-C has 2 parts. Part 1 generates the Symptoms score, and Part 2 generates the Activity and Impacts scores. Total score (0 to 100) is the sum of all scores. Higher scores indicate greater health impairment. Higher score indicate worsening.
EXACT-Respiratory Symptoms (E-RS) | Baseline (for Part 2: participants with chronic obstructive pulmonary disease)
  E-RS is a 11 respiratory system items scoring algorithm to assess the severity of respiratory symptoms in participants with Chronic Obstructive Pulmonary Disease (COPD). Each item has either 5 or 6 response options. Higher score indicate more severe COPD.
Number of participants with adverse events | Up to 1 month (for Part 1: healthy participants and for all Part 2 participants); and Up to 1 year (for Part 1: participants with asthma)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- United States (9):
  - Birmingham, Alabama
  - New Haven, Connecticut
  - Chicago, Illinois
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Galveston, Texas
- Canada (4):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- København NV, Denmark
- France (2):
  - Bordeaux Pessac N/A
  - Marseille
- Germany (2):
  - Frankfurt
  - Lübeck
- Rotterdam, Netherlands
- Bucharest, Romania
- Manchester, United Kingdom

REFERENCES:
- [Derived] Cass SP, Yang Y, Xiao J, McGrath JJC, Fantauzzi MF, Thayaparan D, Wang F, Liang Z, Long F, Stevenson CS, Chen R, Stampfli MR. Current smoking status is associated with reduced sputum immunoglobulin M and G expression in COPD. Eur Respir J. 2021 Feb 4;57(2):1902338. doi: 10.1183/13993003.02338-2019. Print 2021 Feb. No abstract available. PMID 32883677
- [Derived] Loza MJ, Djukanovic R, Chung KF, Horowitz D, Ma K, Branigan P, Barnathan ES, Susulic VS, Silkoff PE, Sterk PJ, Baribaud F; ADEPT (Airways Disease Endotyping for Personalized Therapeutics) and U-BIOPRED (Unbiased Biomarkers for the Prediction of Respiratory Disease Outcome Consortium) investigators. Validated and longitudinally stable asthma phenotypes based on cluster analysis of the ADEPT study. Respir Res. 2016 Dec 15;17(1):165. doi: 10.1186/s12931-016-0482-9. PMID 27978840